CLINICAL TRIAL: NCT04721041
Title: Efficacy and Safety of Washed Microbiota Transplantation for the Treatment of Oncotherapy-Related Intestinal Complications
Brief Title: Washed Microbiota Transplantation for the Treatment of Oncotherapy-Related Intestinal Complications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cancer-CN-202010
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Intestinal Complications; Cancer
Keywords: Fecal Microbiota Transplantation; Washed Microbiota Transplantation; Oncotherapy; Cancer; Intestinal dysbiosis
MeSH Terms: conditions — Neoplasms | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Washed Microbiota Transplantation (WMT) (Experimental): Patients undergo once WMT a day for three consecutive days.
  Interventions: Other: Washed Microbiota Transplantation (WMT)
- Basic treatment (No Intervention): Basic treatment based on the lastest clinical guidelines

INTERVENTIONS:
Other: Washed Microbiota Transplantation (WMT) — Washed microbiota suspension delivered through mid-gut and lower-gut
  Other Names: fecal microbiota transplantation
  Arms: Washed Microbiota Transplantation (WMT)

SUMMARY:
Gut microbiota, known as "unrecognized organs", is closely related to the occurrence and development of tumors. Cancer is thought to occur secondary to local chronic inflammation. And some bacteria, such as Helicobacter pylori, also have direct genotoxicity, changing intracellular signaling pathways and thus causing abnormal cell growth. Systemic intestinal dysbiosis may lead to cancer, and fecal microbiota transplantation (FMT) can be a new weapon in anti-cancer treatment.Washed microbiota transplantation (WMT), a new stage of FMT, is based on the automatic microfiltration machine (GenFMTer, Nanjing, China) and the following repeated centrifugation plus suspension with support from specific facilities. The investigators conducted a prospective, one-arm, open-label study on the efficacy and safety of WMT in the treatment of oncotherapy-related complications. This study aimed to exploring the therapeutic potential of WMT in the treatment of oncotherapy-related intestinal complications and improving the quality of life of patients.

DETAILED DESCRIPTION:
Gut microbiota, known as "unrecognized organs", is closely related to the occurrence and development of tumors. Cancer is thought to occur secondary to local chronic inflammation. And some bacteria, such as Helicobacter pylori, also have direct genotoxicity, changing intracellular signaling pathways and thus causing abnormal cell growth. Systemic intestinal dysbiosis may lead to cancer, and fecal microbiota transplantation (FMT) can be a new weapon in anti-cancer treatment. The reduction of intestinal flora diversity may lead to intestinal dysbiosis, thereby reducing the body immunity and promoting the formation and development of neoplasm. It has been reported that FMT can be used to treat melanoma, liver cancer and prostate cancer after immunotherapy failed. But the mechanism of gut microbiota on the tumor itself remains to be further explored. In 2019, an Italian study reports the efficacy of FMT for diarrhea induced by tyrosine kinase inhibitors in the treatment of renal cell carcinoma, suggesting the therapeutic potential of gut microbiota for tumor-related gastrointestinal complications [1].

Fecal Microbiota transplantation (FMT), the most classic way to treat diseases using gut microbiota [2], refers to the transplantation of functional microbiota in the feces of healthy people into the intestines of patients. It can reconstruct the overall gut microbiota of patients, thus treating gastrointestinal diseases and external gastrointestinal diseases of patients. In 2013, FMT was for the first time coined into the treatment guidelines on recurrent CDI, and now it plays an important role as a key treatment for clostridium difficile infection [3]. Washed microbiota transplantation (WMT), a new stage of FMT, is based on the automatic microfiltration machine (GenFMTer, Nanjing, China) and the following repeated centrifugation plus suspension with support from specific facilities. Compared with manual FMT, WMT can reduce the rate of adverse events (such as fever, diarrhea, abdominal pain, abdominal distension, nausea and vomiting, etc.) without affecting the efficacy. In addition, Zhang et al. have proved that WMT is better than the manual preparation of FMT in improving safety, enriching the precise amount of microbiota and quality controllable in practice [4]. In December 2019, A panel of 28 experts from 22 hospitals or institutes in 15 cities has contributed to the "Nanjing consensus on methodology of washed microbiota transplantation" according to the international standards, and the consensus is published in Chinese Medical Journal in July 2020 [5].

Therefore, the investigators conducted a prospective, one-arm, open-label study on the efficacy and safety of WMT in the treatment of oncotherapy-related intestinal complications. This study aimed to exploring the therapeutic potential of WMT in the treatment of oncotherapy-related intestinal complications and improving the quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old; 2. Diagnosed as malignant tumor; 3. Patients who underwent cancer-related treatment suffering from gastrointestinal symptoms(e.g., abdominal pain, diarrhea, abdominal distension, and difficulty defecating) occurred after standard tumor therapy (such as chemotherapy, radiation, immunotherapy, surgical treatment, etc.); 4. Estimated time of survival ≥ 3 months, and vital signs were stable); 5. Physically qualified and intended to undergo FMT;

Exclusion Criteria:

* 1. Patients who were pregnant or nursing; 2. Patients who were unable or unwilling to undergo a gastroscopy or colonoscopy; 3. Patients with cardiopulmonary failure; 4. Antibiotics, PPI, probiotics, and other drugs that alter gut microbiota were used in the previous week; 5. history of inflammatory bowel disease and intestinal symptoms unrelated to tumor treatment; 6.Serious uncontrolled diseases and acute infectious diseases；

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Scores of gastrointestinal symptoms | 8 weeks
  Gastrointestinal symptoms will be evaluated according to NCI-CTC 5.0
Stool frequency and consistency | 8 weeks
  Stool frequency and consistency will be evaluated according to The Bristol Stool Form Scale (BSFS).

SECONDARY OUTCOMES:
Adverse events | 1 year
  New onset of symptoms and the exacerbation of previous symptoms were recorded as adverse events (AEs)
Karnofsky Performance Status (KPS) scale | 8 weeks
  Changes in functional status of patients will be assessed according to the Karnofsky Performance Status (KPS) scale (ranging from 0 [dead] to 100 [normal activity, no evidence of disease])

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prisciandaro M, Ratta R, Massari F, Fornarini G, Caponnetto S, Iacovelli R, De Giorgi U, Facchini G, Scagliarini S, Sabbatini R, Caserta C, Peverelli G, Mennitto A, Verzoni E, Procopio G. Safety and Efficacy of Cabozantinib for Metastatic Nonclear Renal Cell Carcinoma: Real-world Data From an Italian Managed Access Program. Am J Clin Oncol. 2019 Jan;42(1):42-45. doi: 10.1097/COC.0000000000000478. PMID 30204614
- [Background] Surawicz CM, Brandt LJ, Binion DG, Ananthakrishnan AN, Curry SR, Gilligan PH, McFarland LV, Mellow M, Zuckerbraun BS. Guidelines for diagnosis, treatment, and prevention of Clostridium difficile infections. Am J Gastroenterol. 2013 Apr;108(4):478-98; quiz 499. doi: 10.1038/ajg.2013.4. Epub 2013 Feb 26. PMID 23439232
- [Background] Zhang T, Lu G, Zhao Z, Liu Y, Shen Q, Li P, Chen Y, Yin H, Wang H, Marcella C, Cui B, Cheng L, Ji G, Zhang F. Washed microbiota transplantation vs. manual fecal microbiota transplantation: clinical findings, animal studies and in vitro screening. Protein Cell. 2020 Apr;11(4):251-266. doi: 10.1007/s13238-019-00684-8. Epub 2020 Jan 9. PMID 31919742